CLINICAL TRIAL: NCT02537431
Title: An Open-Label, Single-Arm, Phase 3 Study to Evaluate the Effects of KRN23 on Osteomalacia in Adults With X-linked Hypophosphatemia (XLH)
Brief Title: Open Label Study of KRN23 on Osteomalacia in Adults With X-linked Hypophosphatemia (XLH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX023-CL304
Expanded Access: NCT03775187 (Available)
Record Dates: First submitted 2015-08-25; First posted 2015-09-01 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: X-linked Hypophosphatemia
Keywords: KRN23; Fibroblast growth factor 23 (FGF23); XLH; X-linked Hypophosphatemia
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Open-Label Burosumab Q4W (Experimental): 1.0 mg/kg burosumab monthly (Q4W), calculated based on baseline weight and up to a maximum dose of 90 mg.
  Interventions: Biological: burosumab

INTERVENTIONS:
Biological: burosumab — solution for subcutaneous injection
  Other Names: KRN23; UX023; Crysvita

SUMMARY:
The primary objective of this study is to establish the effect of KRN23 treatment on improvement in XLH-associated osteomalacia as determined by osteoid volume (osteoid volume/bone volume, OV/BV).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 - 65 years, inclusive
2. Diagnosis of XLH supported by classic clinical features of adult XLH (such as short stature or bowed legs), and at least one of the following at Screening:

   * Documented phosphate regulating gene with homology to endopeptidases located on the X chromosome (PHEX) PHEX mutation in either the patient or in a directly related family member with appropriate X-linked inheritance
   * Serum intact FGF23 (iFGF23) level > 30 pg/mL by Kainos assay
3. Biochemical findings consistent with XLH based on overnight fasting (min. 8 hours):

   * Serum phosphorus < 2.5 mg/dL at Screening
   * Ratio of renal tubular maximum phosphate reabsorption rate to glomerular filtration rate (TmP/GFR) < 2.5 mg/dL at Screening
4. Presence of skeletal pain attributed to XLH/osteomalacia, as defined by a score of ≥ 4 on the Brief Pain Inventory question 3 (BPI-Q3, Worst Pain) at Screening. (Skeletal pain that, in the opinion of the investigator, is attributed solely to causes other than XLH/osteomalacia-for example, back pain or joint pain in the presence of severe osteoarthritis by radiograph in that anatomical location-in the absence of any skeletal pain likely attributed to XLH/osteomalacia should not be considered for eligibility)
5. Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min (using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation) or estimated glomerular filtration rate (eGFR) eGFR of 45 to <60 mL/min at Screening with confirmation that the renal insufficiency is not due to nephrocalcinosis
6. Provide written informed consent after the nature of the study has been explained, and prior to any research-related procedures. If the subject in a minor, provide written assent and have a legally authorized representative willing and able to provide written informed consent, after the nature of the study has been explained, and prior to any research-related procedures
7. Willing to provide access to prior medical records for the collection of biochemical and radiographic data and disease history
8. Females of child-bearing potential must have a negative urine pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not to be of childbearing potential include those who have been in menopause for at least two years prior to Screening, or have had tubal ligation at least one year prior to Screening, or have had a total hysterectomy or bilateral salpingo-oophorectomy.
9. Participants of child-bearing potential or with partners of child-bearing potential who have not undergone a total hysterectomy or a bilateral salpingo-oophorectomy and are sexually active must consent to use two effective methods of contraception as determined by the site investigator (i.e. oral hormonal contraceptives, patch hormonal contraceptives, vaginal ring, intrauterine device, physical double-barrier methods, surgical hysterectomy, vasectomy, tubal ligation, or true abstinence) from the period following the signing of the informed consent through 12 weeks after last dose of study drug
10. Must, in the opinion of the investigator, be willing and able to complete all aspects of the study, adhere to the study visit schedule and comply with the assessments

Exclusion Criteria:

1. Use of any pharmacologic vitamin D metabolite or analog (e.g. calcitriol, doxercalciferol, and paricalcitol) within the 2 years before Screening
2. Use of oral phosphate within 2 years before Screening
3. Use of aluminum hydroxide antacids, acetazolamides, and thiazides within 7 days prior to Screening
4. Use of bisphosphonates in the 2 years prior to Screening
5. Use of denosumab in the 6 months prior to Screening
6. Use of teriparatide in the 2 months prior to Screening
7. Chronic use of systemic corticosteroids defined as more than 10 days in the 2 months prior to Screening
8. Corrected serum calcium level ≥ 10.8 mg/dL (2.7 mmol/L) at Screening
9. Serum intact parathyroid hormone (iPTH) ≥ 2.5 times the upper limit of normal (ULN) at Screening
10. Use of medication to suppress parathyroid hormone (PTH) (cinacalcet for example) within 60 days prior to Screening
11. Prothrombin time/Partial thromboplastin time (PT/PTT) outside the normal range at Screening
12. Evidence of any disease or use of anticoagulant medication (such as warfarin, heparin, direct thrombin inhibitors, or Xa inhibitors (xabans) that, in the opinion of the investigator, cannot be discontinued) that may increase the risk of bleeding during the biopsy procedure
13. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study
14. Unable or unwilling to withhold prohibited medications throughout the study
15. Documented dependence on narcotics
16. Use of KRN23, or any other therapeutic monoclonal antibody within 90 days prior to Screening
17. Use of investigational product or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.

    OR, in Japan, use of any investigational product or investigational medical device within 4 months prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
18. Presence or history of any hypersensitivity, allergic or anaphylactic reactions to any monoclonal antibody or KRN23 excipients that, in the judgment of the investigator, places the subject at increased risk for adverse effects
19. History of allergic reaction or adverse reactions to tetracycline or demeclocycline
20. Prior history of positive test for human immunodeficiency virus antibody, hepatitis B surface antigen, and/or hepatitis C antibody
21. History of recurrent infection (other than dental abscesses, which are known to be associated with XLH) or predisposition to infection, or of known immunodeficiency
22. Presence of malignant neoplasm (except basal cell carcinoma)
23. Presence of a concurrent disease or condition that would interfere with study participation or affect safety
24. Presence or history of any condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2018-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - UCSF Medical Center at Mission, San Francisco, California
  - Yale University School of Medicine - Yale New-Haven Hospital/Yale Center for Clinical Investigation, New Haven, Connecticut
  - Indiana University Department of Medicine University Hospital, Indianapolis, Indiana
  - Duke University Medical Center, Durham, North Carolina
  - Houston Methodist Hospital, Houston, Texas
- Canada (2):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Shriners Hospital for Children, Montreal, Quebec
- Aarhus University Hospital-Dept of Endocrinology and Internal Medicine, Aarhus, Denmark
- France (2):
  - CHU de Bicêtre, Service d'Endocrinologie et des Maladies de la Reproduction, Le Kremlin-Bicêtre
  - CHU Paris Centre - Hôpital Cochin, Paris
- Japan (3):
  - Osaka University Hospital, Osaka
  - Hokkaido University Hospital, Sapporo
  - The University of Tokyo Hospital, Tokyo
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Fratzl-Zelman N, Hartmann MA, Gamsjaeger S, Rokidi S, Paschalis EP, Blouin S, Zwerina J. Bone Matrix Mineralization and Response to Burosumab in Adult Patients With X-Linked Hypophosphatemia: Results From the Phase 3, Single-Arm International Trial. J Bone Miner Res. 2022 Sep;37(9):1665-1678. doi: 10.1002/jbmr.4641. Epub 2022 Aug 10. PMID 35775373

RESULTS

PARTICIPANT FLOW:
Period: Open-Label Period (Week 0 to Week 48)
Arm/Group | Open-Label Burosumab Q4W
Started | 14 (Screened and received at least 1 dose of study drug.)
Completed | 13 (Completed Open-Label Period (Week 0 - Week 48))
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Treatment Extension Period I
Arm/Group | Open-Label Burosumab Q4W
Started | 13
Completed | 13
Not Completed | 0
Period: Treatment Extension Period II
Arm/Group | Open-Label Burosumab Q4W
Started | 8 (5 participants completing Treatment Extension Period I did not enter Treatment Extension Period II)
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open-Label Burosumab Q4W: 1.0 mg/kg Q4W, calculated based on baseline weight and up to a maximum dose of 90 mg.
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.13 (8.725)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Osteoid Volume/Bone Volume (OV/BV) [Mean (Standard Deviation); unit: percentage of osteoid volume] — Percent of a given volume of bone tissue that consists of unmineralized bone (osteoid). Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data; participants with non-missing results.
  percentage of osteoid volume
    number analyzed (Participants) | 10
    (all) | 26.12 (12.357)
Serum Phosphorus [Mean (Standard Deviation); unit: mg/dL] | 2.24 (0.396)
Osteoid Thickness (O.Th) [Mean (Standard Deviation); unit: µm] — Mean thickness, given in micrometers, for osteoid seams. Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data.
  µm
    number analyzed (Participants) | 11
    (all) | 17.21 (4.105)
Osteoid Surface/Bone Surface (OS/BS) [Mean (Standard Deviation); unit: percentage of osteoid surface] — Percent of bone surface covered in osteoid. Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data.
  percentage of osteoid surface
    number analyzed (Participants) | 11
    (all) | 91.73 (3.438)
Mineralization Lag Time (MLt) [Mean (Standard Deviation); unit: days] — Average time interval between osteoid formation and its subsequent mineralization; calculated by dividing the osteoid thickness by the adjusted apposition rate (O.Th/Aj.AR). Aj.AR; amount of new bone created (bone formation rate over the entire osteoid surface). The imputed result was used for some of the baseline data for MLt. Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data.
  days
    number analyzed (Participants) | 11
    (all) | 1539.81 (1587.086)
Mineral Apposition Rate (MAR) [Mean (Standard Deviation); unit: µm/day] — Linear rate of new bone deposition; mean distance between the double labels, divided by the time interval between them. Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data.
  µm/day
    number analyzed (Participants) | 11
    (all) | 0.58 (0.448)
Mineralizing Surface/Bone Surface (MS/BS) [Mean (Standard Deviation); unit: percentage of mineralizing surface] — Percent of bone surface that displays a tetracycline label reflecting active mineralization; calculated as the double-labeled surface plus one half of the single-labeled surface and is expressed as a function of total bone surface ([dLS + sLS/2]/BS). It is a measure of the proportion of bone surface upon which new mineralized bone was being deposited during the period of tetracycline labeling. Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data.
  percentage of mineralizing surface
    number analyzed (Participants) | 11
    (all) | 5.99 (4.763)
Bone Formation Rate/Bone Surface (BFR/BS) [Mean (Standard Deviation); unit: µm^3/µm^2/year] — Amount of new bone formed in unit time per unit of bone surface; calculated by multiplying MS/BS by the MAR (see previous measure descriptions for MS/BS and MAR definitions). Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data; participants with non-missing results.
  µm^3/µm^2/year
    number analyzed (Participants) | 6
    (all) | 26.68 (19.480)
Bone Formation Rate/Osteoblast Surface (BFR/OS) [Mean (Standard Deviation); unit: µm^3/µm^2/year] — Bone formation rate to osteoid surface ratio, related to the adjusted apposition rate (Aj.AR; amount of new bone created [bone formation rate over the entire osteoid surface]). Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data; participants with non-missing results.
  µm^3/µm^2/year
    number analyzed (Participants) | 4
    (all) | 2309.00 (2941.970)
Bone Formation Rate/Bone Volume (BFR/BV) [Mean (Standard Deviation); unit: percent/year] — BFR/BV is equivalent to bone turnover rate. Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data; participants with non-missing results.
  percent/year
    number analyzed (Participants) | 6
    (all) | 38.33 (37.173)
1,25(OH) 2D [Mean (Standard Deviation); unit: pg/mL] — Population: Full Analysis Set: enrolled and dosed participants with a baseline measurement.
  pg/mL
    number analyzed (Participants) | 12
    (all) | 37.25 (11.686)
24-Hour Urinary Phosphorus [Mean (Standard Deviation); unit: g/24hr] — Population: Full Analysis Set: enrolled and dosed participants with a baseline measurement.
  g/24hr
    number analyzed (Participants) | 12
    (all) | 0.82 (0.237)
Ratio of Renal Tubular Maximum Reabsorption Rate of Phosphate to Glomerular Filtration Rate(TmP/GFR) [Mean (Standard Deviation); unit: mg/dL] | 1.87 (0.307)
Tubular Reabsorption of Phosphate (TRP) [Mean (Standard Deviation); unit: fraction of phosphorus reabsorbed] | 0.84 (0.048)
Procollagen Type 1 N-Propeptide (P1NP) [Mean (Standard Deviation); unit: ng/mL] | 77.00 (33.273)
Carboxy-Terminal Cross-Linked Telopeptide of Type I Collagen (CTx-I) [Mean (Standard Deviation); unit: pg/mL] | 646.93 (401.641)
Bone-Specific Alkaline Phosphatase (BALP) [Mean (Standard Deviation); unit: μg/L] | 20.43 (9.288)
Mineralizing Surface/OsteoidSurface (MS/OS) [Mean (Standard Deviation); unit: percentage of mineralizing surface] — Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data; participants with non-missing results.
  percentage of mineralizing surface
    number analyzed (Participants) | 11
    (all) | 6.47 (5.120)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in OV/BV at Week 48
Description: OV/BV: percent of a given volume of bone tissue that consists of unmineralized bone (osteoid).
Time Frame: Baseline, 48 weeks
Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data; participants with non-missing results.
Measure: Mean (Standard Deviation); unit: percentage change of unmineralized bone
Groups:
- Open-Label Burosumab Q4W: 1.0 mg/kg burosumab Q4W, calculated based on baseline weight and up to a maximum dose of 90 mg.
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 10
percentage change of unmineralized bone | -54.18 (20.211)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Test type: Other; p < 0.0001, t-test — The null hypothesis of no mean percent change from baseline is tested using t-test; Mean = -54.18, 95% CI 2-sided [-68.64 to -39.72]

2. Secondary Outcome: Percentage of Participants Achieving Mean Serum Phosphorus Levels Above the Lower Limit of Normal (LLN) at the Mid-Point of the Dose Interval, as Averaged Across Dose Cycles Between Baseline and Week 24
Description: The LLN was defined as 2.5 mg/dL (0.81 mmol/L). The 95% confidence interval (CI) was calculated using Wilson score method.
Time Frame: Baseline, up to 24 weeks
Population: Full Analysis Set: all enrolled participants who receive at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
percentage of participants | 92.9 [68.5 to 98.7]
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Test type: Other; p < 0.0001, binomial test — The p-value is for testing the proportion of participants achieving the mean serum phosphorus levels above the LLN (2.5 mg/dL [0.81 mmol/L]) against 0% from the binomial test

3. Secondary Outcome: Percent Change From Baseline in O.Th at Week 48
Description: O.Th: mean thickness, given in micrometers, for osteoid seams.
Time Frame: Baseline, 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change in thickness
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 11
percentage change in thickness | -32.21 (11.966)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Test type: Other; p < 0.0001, t-test — The null hypothesis of no mean percent change from baseline is tested using t-test; Mean = -32.21, 95% CI 2-sided [-40.25 to -24.17]

4. Secondary Outcome: Percent Change From Baseline in OS/BS at Week 48
Description: OS/Bs: percent of bone surface covered in osteoid.
Time Frame: Baseline, 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change of bone surface covered
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 11
percent change of bone surface covered | -26.00 (15.012)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Test type: Other; p = 0.0002, t-test — The null hypothesis of no mean percent change from baseline is tested using t-test; Mean = -26.00, 95% CI 2-sided [-36.08 to -15.91]

5. Secondary Outcome: Percent Change From Baseline in MLt at Week 48
Description: MLt: average time interval between osteoid formation and its subsequent mineralization; calculated by dividing the osteoid thickness by the adjusted apposition rate (O.Th/Aj.AR). Aj.AR; amount of new bone created (bone formation rate over the entire osteoid surface). Based on imputed MLt values.
Time Frame: Baseline, 48 weeks
Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data who had non-missing results.
Measure: Mean (Standard Deviation); unit: percent change in average time interval
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 10
percent change in average time interval | -52.24 (58.487)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Test type: Other; p = 0.0199, t-test — The null hypothesis of no mean percent change from baseline is tested using t-test; Mean = -52.24, 95% CI 2-sided [-94.08 to -10.41]

6. Secondary Outcome: Change From Baseline in MAR at Week 48
Description: MAR: linear rate of new bone deposition; mean distance between the double labels, divided by the time interval between them.
Time Frame: Baseline, 48 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µm/day
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 11
µm/day | 0.04 (0.506)

7. Secondary Outcome: Change From Baseline in MS/BS at Week 48
Description: MS/BS: percent of bone surface that displays a tetracycline label reflecting active mineralization; calculated as the double-labeled surface plus one half of the single-labeled surface and is expressed as a function of total bone surface ([dLS + sLS/2]/BS). It is a measure of the proportion of bone surface upon which new mineralized bone was being deposited during the period of tetracycline labeling.
Time Frame: Baseline, 48 weeks
Population: Primary Analysis Set: enrolled participants with baseline and follow-up (Week 48/end of treatment) bone biopsy data who had non-missing data.
Measure: Mean (Standard Deviation); unit: percent of mineralizing surface
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 10
percent of mineralizing surface | 1.32 (4.365)

8. Secondary Outcome: Change From Baseline in BFR/BS at Week 48
Description: BFR/BS: amount of new bone formed in unit time per unit of bone surface; calculated by multiplying MS/BS by the MAR.
  MS/BS: percent of bone surface that displays a tetracycline label reflecting active mineralization; calculated as the double-labeled surface plus one half of the single-labeled surface and is expressed as a function of total bone surface ([dLS + sLS/2]/BS). It is a measure of the proportion of bone surface upon which new mineralized bone was being deposited during the period of tetracycline labeling. MAR: linear rate of new bone deposition; mean distance between the double labels, divided by the time interval between them.
Time Frame: Baseline, 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µm^3/µm^2/year
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 6
µm^3/µm^2/year | -4.90 (27.356)

9. Secondary Outcome: Change From Baseline in BFR/OS at Week 48
Description: BFR/OS: bone formation rate to osteoid surface ratio, related to the Aj.AR (amount of new bone created [bone formation rate over the entire osteoid surface]).
Time Frame: Baseline, 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µm^3/µm^2/year
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 4
µm^3/µm^2/year | -1557.25 (3139.075)

10. Secondary Outcome: Change From Baseline in BFR/BV at Week 48
Description: BFR/BV: equivalent to bone turnover rate.
Time Frame: Baseline, 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of bone turnover/year
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 6
percentage of bone turnover/year | -13.50 (32.904)

11. Secondary Outcome: Percentage of Participants Achieving Mean Serum Phosphorus Levels Above the LLN at the End of the Dosing Cycle Between Baseline and Week 24
Description: The LLN was defined as 2.5 mg/dL (0.81 mmol/L). The 95% CI was calculated using Wilson score method.
Time Frame: Baseline, up to 24 weeks
Population: Full Analysis Set: all enrolled participants who receive at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
percentage of participants | 78.6 [52.4 to 92.4]

12. Secondary Outcome: Mean Change of Serum Phosphorus Levels at the Mid-Point of Dosing Cycle, as Averaged Across Dose Cycles Between Baseline and Week 24
Time Frame: Baseline, up to 24 weeks
Population: Full Analysis Set: all enrolled participants who receive at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
mg/dL | 1.07 (0.300)

13. Secondary Outcome: Percent Change of Serum Phosphorus Levels at the Mid-Point of Dosing Cycle, as Averaged Across Dose Cycles Between Baseline and Week 24
Time Frame: Baseline, up to 24 weeks
Population: Full Analysis Set: all enrolled participants who receive at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: percent change of serum phosphorus level
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
percent change of serum phosphorus level | 50.39 (19.942)

14. Secondary Outcome: Mean Change of Serum Phosphorus Levels at the End of Dosing Cycle, as Averaged Across Dose Cycles Between Baseline and Week 24
Time Frame: Baseline, up to 24 weeks
Population: Full Analysis Set: all enrolled participants who receive at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
mg/dL | 0.46 (0.303)

15. Secondary Outcome: Percentage Change of Serum Phosphorus Levels at the End of Dosing Cycle, as Averaged Across Dose Cycles Between Baseline and Week 24
Time Frame: Baseline, up to 24 weeks
Population: Full Analysis Set: all enrolled participants who receive at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: percent change of serum phosphorus level
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
percent change of serum phosphorus level | 23.32 (19.836)

16. Secondary Outcome: Time-Adjusted Area Under the Curve (AUC) of Serum Phosphorus Between Baseline and Week 24
Time Frame: Baseline, up to 24 weeks
Population: Full Analysis Set: all enrolled participants who receive at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
mg/dL | 3.023 (0.2716)

17. Secondary Outcome: Change From Baseline Over Time in Serum 1,25(OH)2D
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 20, Week 21, Week 22, Week 24, Week 48, Week 60, Week 70, Week 72, Week 84, Week 94, Week 96, Week 108, Week 120, Week 132
Population: Full Analysis Set: all enrolled participants who receive at least one dose of study drug with non-missing results at given time point.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 12
pg/mL
  Week 1 | 107.75 (15.964)
  Week 2 | 48.41 (7.397)
  Week 4 | 13.58 (3.435)
  Week 20 | -1.34 (3.617)
  Week 21 | 31.75 (5.233)
  Week 22: number analyzed (Participants) | 11
  Week 22 | 11.50 (4.060)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -3.04 (4.891)
  Week 48: number analyzed (Participants) | 11
  Week 48 | -1.72 (4.190)
  Week 60: number analyzed (Participants) | 11
  Week 60 | -5.73 (3.395)
  Week 70: number analyzed (Participants) | 11
  Week 70 | 3.36 (3.987)
  Week 72: number analyzed (Participants) | 11
  Week 72 | -5.55 (2.895)
  Week 84: number analyzed (Participants) | 11
  Week 84 | -5.55 (2.962)
  Week 94: number analyzed (Participants) | 11
  Week 94 | 9.63 (4.239)
  Week 96: number analyzed (Participants) | 11
  Week 96 | -6.09 (2.403)
  Week 108: number analyzed (Participants) | 7
  Week 108 | 0.02 (4.714)
  Week 120: number analyzed (Participants) | 2
  Week 120 | 1.45 (4.197)
  Week 132: number analyzed (Participants) | 1
  Week 132 | -1.69 (1.993)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Week 1; Test type: Other; Least Squares Mean (GEE) = 107.75, 95% CI 2-sided [76.46 to 139.03] — From the generalized estimation equation (GEE) model which includes change from baseline for 1, 25 (OH)2 D as the dependent variable, visit as fixed factors, and baseline of 1, 25 (OH)2 D as a covariate, with compound symmetry covariance structure
Statistical Analysis 2: Comparison: Open-Label Burosumab Q4W; Week 2; Test type: Other; LS Mean = 48.41, 95% CI 2-sided [33.91 to 62.91] — From the GEE model which includes the change from baseline for 1, 25 (OH)2 D as the dependent variable, visit as fixed factors, and baseline of 1, 25 (OH)2 D as a covariate, with compound symmetry covariance structure
Statistical Analysis 3: Comparison: Open-Label Burosumab Q4W; Week 4; Test type: Other; LS Mean = 13.58, 95% CI 2-sided [6.85 to 20.31] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 4: Comparison: Open-Label Burosumab Q4W; Week 20; Test type: Other; LS Mean = -1.34, 95% CI 2-sided [-8.43 to 5.75] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 5: Comparison: Open-Label Burosumab Q4W; Week 21; Test type: Other; LS Mean = 31.75, 95% CI 2-sided [21.49 to 42.00] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 6: Comparison: Open-Label Burosumab Q4W; Week 22; Test type: Other; LS Mean = 11.50, 95% CI 2-sided [3.54 to 19.46] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 7: Comparison: Open-Label Burosumab Q4W; Week 24; Test type: Other; LS Mean = -3.04, 95% CI 2-sided [-12.62 to 6.55] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 8: Comparison: Open-Label Burosumab Q4W; Week 48; Test type: Other; p = 0.6821, GEE model; LS Mean = -1.72, 95% CI 2-sided [-9.93 to 6.50] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 9: Comparison: Open-Label Burosumab Q4W; Week 60; Test type: Other; LS mean = -5.73, 95% CI 2-sided [-12.38 to 0.92] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 10: Comparison: Open-Label Burosumab Q4W; Week 70; Test type: Other; LS mean = 3.36, 95% CI 2-sided [-4.45 to 11.18] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 11: Comparison: Open-Label Burosumab Q4W; Week 72; Test type: Other; LS mean = -5.55, 95% CI 2-sided [-11.22 to 0.13] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 12: Comparison: Open-Label Burosumab Q4W; Week 84; Test type: Other; LS mean = -5.55, 95% CI 2-sided [-11.35 to 0.26] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 13: Comparison: Open-Label Burosumab Q4W; Week 94; Test type: Other; LS mean = 9.63, 95% CI 2-sided [1.33 to 17.94] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 14: Comparison: Open-Label Burosumab Q4W; Week 96; Test type: Other; LS mean = -6.09, 95% CI 2-sided [-10.80 to -1.38]
Statistical Analysis 15: Comparison: Open-Label Burosumab Q4W; Week 108; Test type: Other; LS mean = 0.02, 95% CI 2-sided [-9.22 to 9.26] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 16: Comparison: Open-Label Burosumab Q4W; Week 120; Test type: Other; LS mean = 1.45, 95% CI 2-sided [-6.77 to 9.68] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 17: Comparison: Open-Label Burosumab Q4W; Week 132; Test type: Other; LS mean = -1.69, 95% CI 2-sided [-5.60 to 2.21] — [estimate comment as in outcome 17, analysis 2]

18. Secondary Outcome: Change From Baseline Over Time in 24-Hour Urinary Phosphorus
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, Week 72, Week 96, End of Study II (EOSII) (up to Week 141)
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: g/24 hours
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 12
g/24 hours
  Week 12: number analyzed (Participants) | 11
  Week 12 | 0.10 (0.128)
  Week 24 | -0.04 (0.075)
  Week 36 | -0.01 (0.059)
  Week 48: number analyzed (Participants) | 11
  Week 48 | -0.04 (0.076)
  Week 72: number analyzed (Participants) | 11
  Week 72 | 0.00 (0.096)
  Week 96: number analyzed (Participants) | 9
  Week 96 | -0.13 (0.082)
  EOSII: number analyzed (Participants) | 5
  EOSII | -0.07 (0.171)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Week 12; Test type: Other; LS Mean = 0.10, 95% CI 2-sided [-0.15 to 0.35] — From the GEE model; includes change from baseline from baseline for 24-Hour urinary phosphorus as the dependent variable, visit as fixed factors, and baseline of 24-Hour urinary phosphorus as a covariate, with compound symmetry covariance structure
Statistical Analysis 2: Comparison: Open-Label Burosumab Q4W; Week 24; Test type: Other; LS Mean = -0.04, 95% CI 2-sided [-0.19 to 0.11] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 3: Comparison: Open-Label Burosumab Q4W; Week 36; Test type: Other; LS Mean = -0.01, 95% CI 2-sided [-0.12 to 0.11] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 4: Comparison: Open-Label Burosumab Q4W; Week 48; Test type: Other; p = 0.6021, GEE model; LS Mean = -0.04, 95% CI 2-sided [-0.19 to 0.11] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 5: Comparison: Open-Label Burosumab Q4W; Week 72; Test type: Other; LS mean = 0.00, 95% CI 2-sided [-0.19 to 0.19] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 6: Comparison: Open-Label Burosumab Q4W; Week 96; Test type: Other; LS mean = -0.13, 95% CI 2-sided [-0.29 to 0.03] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 7: Comparison: Open-Label Burosumab Q4W; EOS II; Test type: Other; LS mean = -0.07, 95% CI 2-sided [-0.41 to 0.26] — [estimate comment as in outcome 18, analysis 1]

19. Secondary Outcome: Change From Baseline Over Time in TmP/GFR
Description: TmP/GFR: ratio of renal tubular maximum reabsorption rate of phosphate to glomerular filtration rate.
Time Frame: Baseline, Week 2, Week 4, Week 12, Week 22, Week 24, Week 48, Week 60, Week 72, Week 84, Week 96, EOSII (up to Week 141)
Population: Full Analysis Set: all enrolled participants who receive at least one dose of study drug, with non-missing results at given time point.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 13
mg/dL
  Week 2 | 1.76 (0.136)
  Week 4 | 0.78 (0.097)
  Week 12 | 0.58 (0.122)
  Week 22 | 0.87 (0.064)
  Week 24 | 0.44 (0.101)
  Week 48 | 0.20 (0.097)
  Week 60 | 0.30 (0.171)
  Week 72: number analyzed (Participants) | 12
  Week 72 | 0.28 (0.127)
  Week 84 | 0.39 (0.136)
  Week 96 | 0.29 (0.097)
  EOSII: number analyzed (Participants) | 8
  EOSII | 0.21 (0.068)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Week 2; Test type: Other; LS Mean = 1.76, 95% CI 2-sided [1.49 to 2.03] — From the GEE model, which includes the change from baseline for TmP/GFR as the dependent variable, visit as fixed factors, and baseline of TmP/GFR as a covariate, with compound symmetry covariance structure
Statistical Analysis 2: Comparison: Open-Label Burosumab Q4W; Week 4; Test type: Other; LS Mean = 0.78, 95% CI 2-sided [0.59 to 0.97] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 3: Comparison: Open-Label Burosumab Q4W; Week 12; Test type: Other; LS Mean = 0.58, 95% CI 2-sided [0.34 to 0.82] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 4: Comparison: Open-Label Burosumab Q4W; Week 22; Test type: Other; LS Mean = 0.87, 95% CI 2-sided [0.74 to 0.99] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 5: Comparison: Open-Label Burosumab Q4W; Week 24; Test type: Other; LS Mean = 0.44, 95% CI 2-sided [0.24 to 0.64] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 6: Comparison: Open-Label Burosumab Q4W; Week 48; Test type: Other; p = 0.0430, GEE model; LS Mean = 0.20, 95% CI 2-sided [0.01 to 0.38] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 7: Comparison: Open-Label Burosumab Q4W; Week 60; Test type: Other; LS mean = 0.30, 95% CI 2-sided [-0.04 to 0.64] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 8: Comparison: Open-Label Burosumab Q4W; Week 72; Test type: Other; LS mean = 0.28, 95% CI 2-sided [0.03 to 0.52] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 9: Comparison: Open-Label Burosumab Q4W; Week 84; Test type: Other; LS mean = 0.39, 95% CI 2-sided [0.13 to 0.66] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 10: Comparison: Open-Label Burosumab Q4W; Week 96; Test type: Other; LS mean = 0.29, 95% CI 2-sided [0.10 to 0.48] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 11: Comparison: Open-Label Burosumab Q4W; EOSII; Test type: Other; LS mean = 0.21, 95% CI 2-sided [0.08 to 0.34] — [estimate comment as in outcome 19, analysis 1]

20. Secondary Outcome: Change From Baseline Over Time in TRP
Description: TRP: tubular reabsorption of phosphate.
Time Frame: as for outcome 19
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: fraction of phosphorus reabsorbed
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
fraction of phosphorus reabsorbed
  Week 2 | 0.07 (0.005)
  Week 4 | 0.03 (0.013)
  Week 12: number analyzed (Participants) | 13
  Week 12 | 0.01 (0.013)
  Week 22: number analyzed (Participants) | 12
  Week 22 | 0.04 (0.007)
  Week 24 | 0.01 (0.015)
  Week 48: number analyzed (Participants) | 13
  Week 48 | -0.00 (0.021)
  Week 60: number analyzed (Participants) | 13
  Week 60 | 0.03 (0.016)
  Week 72: number analyzed (Participants) | 13
  Week 72 | -0.02 (0.035)
  Week 84: number analyzed (Participants) | 13
  Week 84 | 0.02 (0.019)
  Week 96: number analyzed (Participants) | 13
  Week 96 | 0.02 (0.014)
  EOSII: number analyzed (Participants) | 8
  EOSII | 0.01 (0.011)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Week 2; Test type: Other; LS Mean = 0.07, 95% CI 2-sided [0.06 to 0.08] — From the GEE model, which includes the change from baseline or percent change from baseline for TRP as the dependent variable, visit as fixed factors, and baseline of TRP as a covariate, with compound symmetry covariance structure
Statistical Analysis 2: Comparison: Open-Label Burosumab Q4W; Week 4; Test type: Other; LS Mean = 0.03, 95% CI 2-sided [0.01 to 0.06] — From the GEE model which includes the change from baseline or percent change from baseline for TRP as the dependent variable, visit as fixed factors, and baseline of TRP as a covariate, with compound symmetry covariance structure
Statistical Analysis 3: Comparison: Open-Label Burosumab Q4W; Week 12; Test type: Other; LS Mean = 0.01, 95% CI 2-sided [-0.01 to 0.04] — [estimate comment as in outcome 20, analysis 2]
Statistical Analysis 4: Comparison: Open-Label Burosumab Q4W; Week 22; Test type: Other; LS Mean = 0.04, 95% CI 2-sided [0.02 to 0.05] — [estimate comment as in outcome 20, analysis 2]
Statistical Analysis 5: Comparison: Open-Label Burosumab Q4W; Week 24; Test type: Other; LS Mean = 0.01, 95% CI 2-sided [-0.02 to 0.04]
Statistical Analysis 6: Comparison: Open-Label Burosumab Q4W; Week 48; Test type: Other; p = 0.8377, GEE model; LS Mean = -0.00, 95% CI 2-sided [-0.05 to 0.04] — [estimate comment as in outcome 20, analysis 2]
Statistical Analysis 7: Comparison: Open-Label Burosumab Q4W; Week 60; Test type: Other; LS mean = 0.03, 95% CI 2-sided [-0.00 to 0.06] — [estimate comment as in outcome 20, analysis 2]
Statistical Analysis 8: Comparison: Open-Label Burosumab Q4W; Week 72; Test type: Other; LS mean = -0.02, 95% CI 2-sided [-0.09 to 0.05] — [estimate comment as in outcome 20, analysis 2]
Statistical Analysis 9: Comparison: Open-Label Burosumab Q4W; Week 84; Test type: Other; LS mean = 0.02, 95% CI 2-sided [-0.01 to 0.06] — [estimate comment as in outcome 20, analysis 2]
Statistical Analysis 10: Comparison: Open-Label Burosumab Q4W; Week 96; Test type: Other; LS mean = 0.02, 95% CI 2-sided [-0.01 to 0.05] — [estimate comment as in outcome 20, analysis 2]
Statistical Analysis 11: Comparison: Open-Label Burosumab Q4W; EOSII; Test type: Other; LS mean = 0.01, 95% CI 2-sided [-0.01 to 0.03] — [estimate comment as in outcome 20, analysis 2]

21. Secondary Outcome: Change From Baseline Over Time in P1NP
Description: P1NP: procollagen type 1 N-propeptide.
Time Frame: Baseline, Week 12, Week 24, Week 48, Week 72, Week 96, EOSII (up to Week 141)
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
ng/mL
  Week 12: number analyzed (Participants) | 13
  Week 12 | 99.18 (11.403)
  Week 24 | 104.33 (11.153)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 52.49 (11.554)
  Week 72: number analyzed (Participants) | 13
  Week 72 | 37.29 (12.294)
  Week 96: number analyzed (Participants) | 13
  Week 96 | 29.29 (13.321)
  EOSII: number analyzed (Participants) | 8
  EOSII | 2.14 (10.105)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Week 12; Test type: Other; LS Mean = 99.18, 95% CI 2-sided [76.83 to 121.53] — From the GEE model, which includes the change from baseline for P1NP as the dependent variable, visit as fixed factors, and baseline of P1NP as a covariate, with compound symmetry covariance structure
Statistical Analysis 2: Comparison: Open-Label Burosumab Q4W; Week 24; Test type: Other; LS Mean = 104.33, 95% CI 2-sided [82.47 to 126.19] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Open-Label Burosumab Q4W; Week 48; Test type: Other; p < 0.0001, GEE model; LS Mean = 52.49, 95% CI 2-sided [29.84 to 75.13] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Open-Label Burosumab Q4W; Week 72; Test type: Other; LS mean = 37.29, 95% CI 2-sided [13.19 to 61.38] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 5: Comparison: Open-Label Burosumab Q4W; Week 96; Test type: Other; LS mean = 29.29, 95% CI 2-sided [3.18 to 55.40] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 6: Comparison: Open-Label Burosumab Q4W; EOSII; Test type: Other; LS mean = 2.14, 95% CI 2-sided [-17.67 to 21.94] — [estimate comment as in outcome 21, analysis 1]

22. Secondary Outcome: Percent Change From Baseline Over Time in P1NP
Time Frame: Baseline, Week 12, Week 24, Week 48, Week 72, Week 96, EOSII (up to Week 141)
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: percent change in P1NP
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
percent change in P1NP
  Week 12: number analyzed (Participants) | 13
  Week 12 | 133.08 (13.680)
  Week 24 | 137.80 (15.741)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 76.86 (14.114)
  Week 72: number analyzed (Participants) | 13
  Week 72 | 50.46 (13.659)
  Week 96: number analyzed (Participants) | 13
  Week 96 | 41.36 (11.566)
  EOSII: number analyzed (Participants) | 8
  EOSII | 26.20 (9.919)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Week 12; Test type: Other; LS Mean = 133.08, 95% CI 2-sided [106.26 to 159.89] — From the GEE model, which includes the percent change from baseline for P1NP as the dependent variable, visit as fixed factors, and baseline of P1NP as a covariate, with compound symmetry covariance structure
Statistical Analysis 2: Comparison: Open-Label Burosumab Q4W; Week 24; Test type: Other; LS Mean = 137.80, 95% CI 2-sided [106.95 to 168.65] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 3: Comparison: Open-Label Burosumab Q4W; Week 48; Test type: Other; p < 0.0001, GEE model; LS Mean = 76.86, 95% CI 2-sided [49.20 to 104.53] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 4: Comparison: Open-Label Burosumab Q4W; Week 72; Test type: Other; LS mean = 50.46, 95% CI 2-sided [23.69 to 77.23] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 5: Comparison: Open-Label Burosumab Q4W; Week 96; Test type: Other; LS mean = 41.36, 95% CI 2-sided [18.69 to 64.03] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 6: Comparison: Open-Label Burosumab Q4W; EOSII; Test type: Other; LS mean = 26.20, 95% CI 2-sided [6.76 to 45.64] — [estimate comment as in outcome 22, analysis 1]

23. Secondary Outcome: Change From Baseline Over Time in CTx
Description: CTx: carboxy-terminal cross-linked telopeptide of type I collagen.
Time Frame: Baseline, Week 12, Week 24, Week 48, Week 72, Week 96, EOSII (up to Week 141)
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
pg/mL
  Week 12 | 464.84 (61.696)
  Week 24 | 404.13 (55.948)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 175.13 (44.022)
  Week 72: number analyzed (Participants) | 13
  Week 72 | 143.11 (92.503)
  Week 96: number analyzed (Participants) | 13
  Week 96 | 76.80 (57.357)
  EOSII: number analyzed (Participants) | 8
  EOSII | -41.32 (83.144)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Week 12; Test type: Other; LS Mean = 464.84, 95% CI 2-sided [343.92 to 585.77] — From the GEE model which includes the change from baseline for CTx as the dependent variable, visit as fixed factors, and baseline of CTx as a covariate, with compound symmetry covariance structure
Statistical Analysis 2: Comparison: Open-Label Burosumab Q4W; Week 24; Test type: Other; LS Mean = 404.13, 95% CI 2-sided [294.47 to 513.78] — [estimate comment as in outcome 23, analysis 1]
Statistical Analysis 3: Comparison: Open-Label Burosumab Q4W; Week 48; Test type: Other; p < 0.0001, GEE model; LS Mean = 175.13, 95% CI 2-sided [88.85 to 261.41] — [estimate comment as in outcome 23, analysis 1]
Statistical Analysis 4: Comparison: Open-Label Burosumab Q4W; Week 72; Test type: Other; LS mean = 143.11, 95% CI 2-sided [-38.20 to 324.41] — [estimate comment as in outcome 23, analysis 1]
Statistical Analysis 5: Comparison: Open-Label Burosumab Q4W; Week 96; Test type: Other; LS mean = 76.80, 95% CI 2-sided [-35.62 to 189.22] — [estimate comment as in outcome 23, analysis 1]
Statistical Analysis 6: Comparison: Open-Label Burosumab Q4W; EOSII; Test type: Other; LS mean = -41.32, 95% CI 2-sided [-204.28 to 121.64] — [estimate comment as in outcome 23, analysis 1]

24. Secondary Outcome: Percent Change From Baseline Over Time in CTx
Description: CTx: carboxy-terminal cross-linked telopeptide of type I collagen.
Time Frame: Baseline, Week 12, Week 24, Week 48, Week 72, Week 96, EOSII (up to Week 141)
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: percent change in CTx
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 14
percent change in CTx
  Week 12 | 89.68 (13.316)
  Week 24 | 70.17 (10.341)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 35.86 (7.396)
  Week 72: number analyzed (Participants) | 13
  Week 72 | 34.00 (14.016)
  Week 96: number analyzed (Participants) | 13
  Week 96 | 25.86 (8.461)
  EOSII: number analyzed (Participants) | 8
  EOSII | 17.88 (9.284)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Week 12; Test type: Other; LS Mean = 89.68, 95% CI 2-sided [63.58 to 115.78] — From the GEE model which includes the percent change from baseline for CTx as the dependent variable, visit as fixed factors, and baseline of CTx as a covariate, with compound symmetry covariance structure
Statistical Analysis 2: Comparison: Open-Label Burosumab Q4W; Week 24; Test type: Other; LS Mean = 70.17, 95% CI 2-sided [49.90 to 90.44] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 3: Comparison: Open-Label Burosumab Q4W; Week 48; Test type: Other; p < 0.0001, GEE model; LS Mean = 35.86, 95% CI 2-sided [21.37 to 50.36] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 4: Comparison: Open-Label Burosumab Q4W; Week 72; Test type: Other; LS mean = 34.00, 95% CI 2-sided [6.53 to 61.47] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 5: Comparison: Open-Label Burosumab Q4W; Week 96; Test type: Other; LS mean = 25.86, 95% CI 2-sided [9.27 to 42.44] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 6: Comparison: Open-Label Burosumab Q4W; EOSII; Test type: Other; LS mean = 17.88, 95% CI 2-sided [-0.32 to 36.07] — [estimate comment as in outcome 24, analysis 1]

25. Secondary Outcome: Change From Baseline Over Time in BALP
Description: BALP: bone-specific alkaline phosphatase.
Time Frame: Baseline, Week 12, Week 24, Week 48, Week 72, Week 96, EOSII (up to Week 141)
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: μg/L
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 13
μg/L
  Week 12 | 10.93 (3.547)
  Week 24 | 5.82 (2.980)
  Week 48 | 4.50 (3.990)
  Week 72: number analyzed (Participants) | 12
  Week 72 | 3.13 (2.435)
  Week 96 | 1.14 (2.028)
  EOSII: number analyzed (Participants) | 8
  EOSII | -5.80 (3.396)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Week 12; Test type: Other; LS Mean = 10.93, 95% CI 2-sided [3.98 to 17.89] — From the GEE model, which includes the change from baseline for Bone ALP as the dependent variable, visit as fixed factors, and baseline of Bone ALP as a covariate, with compound symmetry covariance structure
Statistical Analysis 2: Comparison: Open-Label Burosumab Q4W; Week 24; Test type: Other; LS Mean = 5.82, 95% CI 2-sided [-0.02 to 11.66] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Open-Label Burosumab Q4W; Week 48; Test type: Other; p = 0.2592, GEE model; LS Mean = 4.50, 95% CI 2-sided [-3.32 to 12.32] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Open-Label Burosumab Q4W; Week 72; Test type: Other; LS mean = 3.13, 95% CI 2-sided [-1.64 to 7.90] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Open-Label Burosumab Q4W; Week 96; Test type: Other; LS mean = 1.14, 95% CI 2-sided [-2.84 to 5.11] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Open-Label Burosumab Q4W; EOSII; Test type: Other; LS mean = -5.80, 95% CI 2-sided [-12.46 to 0.85] — [estimate comment as in outcome 25, analysis 1]

26. Secondary Outcome: Percent Change From Baseline Over Time in BALP
Description: BALP: bone-specific alkaline phosphatase.
Time Frame: Baseline, Week 12, Week 24, Week 48, Week 72, Week 96, EOSII (up to Week 141)
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: percent change in BALP
Arm/Group | Open-Label Burosumab Q4W
Number analyzed (Participants) | 13
percent change in BALP
  Week 12 | 52.54 (15.999)
  Week 24 | 31.37 (11.808)
  Week 48 | 24.35 (17.630)
  Week 72: number analyzed (Participants) | 12
  Week 72 | 15.13 (13.431)
  Week 96 | 6.92 (10.387)
  EOSII: number analyzed (Participants) | 8
  EOSII | -27.30 (12.767)
Statistical Analysis 1: Comparison: Open-Label Burosumab Q4W; Week 12; Test type: Other; LS Mean = 52.54, 95% CI 2-sided [21.18 to 83.90] — From the GEE model, which includes the percent change from baseline for Bone ALP as the dependent variable, visit as fixed factors, and baseline of Bone ALP as a covariate, with compound symmetry covariance structure
Statistical Analysis 2: Comparison: Open-Label Burosumab Q4W; Week 24; Test type: Other; LS Mean = 31.37, 95% CI 2-sided [8.23 to 54.51] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 3: Comparison: Open-Label Burosumab Q4W; Week 48; Test type: Other; p = 0.1672, GEE model; l = 24.35, 95% CI 2-sided [-10.20 to 58.90] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 4: Comparison: Open-Label Burosumab Q4W; Week 72; Test type: Other; LS mean = 15.13, 95% CI 2-sided [-11.19 to 41.46] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 5: Comparison: Open-Label Burosumab Q4W; Week 96; Test type: Other; LS mean = 6.92, 95% CI 2-sided [-13.44 to 27.28] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 6: Comparison: Open-Label Burosumab Q4W; EOSII; Test type: Other; LS mean = -27.30, 95% CI 2-sided [-52.33 to -2.28] — [estimate comment as in outcome 26, analysis 1]

ADVERSE EVENTS:
Time Frame: Week 0 to EOSII (up to Week 141). Mean (SE) duration of exposure to study drug was 716 (35.1) days
Description: Treatment-emergent adverse events are presented.
Arm/Group | Open-Label Burosumab Q4W
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 4/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Burosumab Q4W (N=14)
Atrial Fibrillation (Cardiac disorders) | 1
Obstruction Gastric (Gastrointestinal disorders) | 1
Splenic Rupture (Injury, poisoning and procedural complications) | 1
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Burosumab Q4W (N=14)
Bradycardia (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Abdominal Discomfort (Gastrointestinal disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2
Gingival Pain (Gastrointestinal disorders) | 1
Gingival Swelling (Gastrointestinal disorders) | 2
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1
Mouth Ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oral Pain (Gastrointestinal disorders) | 1
Periodontal Disease (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Vomiting Projectile (Gastrointestinal disorders) | 1
Application Site Rash (General disorders) | 1
Asthenia (General disorders) | 2
Chest Discomfort (General disorders) | 2
Chest Pain (General disorders) | 1
Drug Withdrawal Syndrome (General disorders) | 1
Fatigue (General disorders) | 3
Influenza Like Illness (General disorders) | 2
Injection Site Bruising (General disorders) | 1
Injection Site Pain (General disorders) | 2
Injection Site Pruritus (General disorders) | 1
Injection Site Reaction (General disorders) | 2
Injection Site Urticaria (General disorders) | 3
Local Swelling (General disorders) | 1
Nodule (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Pain (General disorders) | 5
Peripheral Swelling (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatic Steatosis (Hepatobiliary disorders) | 1
Drug Hypersensitivity (Immune system disorders) | 2
Seasonal Allergy (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Conjunctivitis Bacterial (Infections and infestations) | 1
Gingival Abscess (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Influenza (Infections and infestations) | 4
Laryngitis (Infections and infestations) | 1
Lice Infestation (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Periodontitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pharyngitis Streptococcal (Infections and infestations) | 2
Postoperative Wound Infection (Infections and infestations) | 1
Respiratory Tract Infection Viral (Infections and infestations) | 1
Root Canal Infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Tooth Abscess (Infections and infestations) | 7
Tooth Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Vulvovaginal Mycotic Infection (Infections and infestations) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Incision Site Pruritus (Injury, poisoning and procedural complications) | 2
Injection Related Reaction (Injury, poisoning and procedural complications) | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1
Post Procedural Swelling (Injury, poisoning and procedural complications) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 7
Stress Fracture (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 2
Tooth Injury (Injury, poisoning and procedural complications) | 1
Blood 25-Hydroxycholecalciferol Decreased (Investigations) | 2
Blood Calcium Decreased (Investigations) | 1
Blood Cholesterol Increased (Investigations) | 1
Blood Glucose Increased (Investigations) | 1
Blood Parathyroid Hormone Increased (Investigations) | 1
Blood Pressure Increased (Investigations) | 1
Blood Testosterone Decreased (Investigations) | 1
Blood Uric Acid Increased (Investigations) | 1
Ejection Fraction Decreased (Investigations) | 1
Eosinophil Count Increased (Investigations) | 1
Ultrasound Kidney Abnormal (Investigations) | 1
Vitamin D Decreased (Investigations) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 6
Bone Pain (Musculoskeletal and connective tissue disorders) | 3
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Joint Instability (Musculoskeletal and connective tissue disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1
Spinal Pain (Musculoskeletal and connective tissue disorders) | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Amnesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysaesthesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 3
Migraine (Nervous system disorders) | 1
Motor Dysfunction (Nervous system disorders) | 1
Nerve Compression (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 3
Restless Legs Syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 4
Confusional State (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Depressive Symptom (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Irritability (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Glycosuria (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1
Uterine Haemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 4
Sinus Perforation (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Skin Irritation (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Xanthoma (Skin and subcutaneous tissue disorders) | 2
Hot Flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT02537431/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT02537431/SAP_001.pdf